CLINICAL TRIAL: NCT05228626
Title: Safety and Efficacy of COVIDEX™ Therapy in Management of Adult Covid-19 Patients in Uganda: A Randomized Double-blind Placebo Controlled Adaptive Phase 2 B Clinical Trial.
Brief Title: Safety and Efficacy of COVIDEX™ Therapy in Management of Adult COVID-19 Patients in Uganda.
Acronym: COT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Associate professor, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBS-2022-129
Record Dates: First submitted 2022-02-07; First posted 2022-02-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: COVIDEX
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to two trial arms. Arm1: the control arm will be composed of Standard of care for treating COVID-19 in Uganda as recommended by the ministry of Health plus the Placebo Arm 2: the Intervention arm will be composed of the intervention plus the standard of care for treating COVID-19 in Uganda as recommended by the ministry of Health
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the participant and study clinicians and other data collectors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care plus placebo arm (Placebo Comparator): Will contain standard of care plus placebo
  Interventions: Drug: COVIDEX
- Stanadard of care plus COVIDEX arm (Experimental): Will contain the standard of care plus the intervention given for 3 times daily for seven days
  Interventions: Drug: COVIDEX

INTERVENTIONS:
Drug: COVIDEX — COVIDEXTm is a prepared plant extract of Zanthoxylum and Warbugia species that is reported to have antiviral agents, one of which berberine with in vitro activity against SARS COV-2, the causative agent for COVID-19 disease. Others constituents in COVIDEX include alkaloids, sponins, reducing sugars and acidic compounds. IT is given either 2 drops nasally plus 6 drops orally or 6 oral drops only of COVIDEXTm three times daily for 7 days.

SUMMARY:
The SARS-CoV-2 pandemic continues to grow, with over 350,000 new infections and over 7,000 daily global deaths in May 2021 (WHO, 2021a). The current supplies of protective vaccines are too low to cover the worldwide demand hence researchers worldwide are urgently looking for interventions to prevent new infections, prevent disease progression, and lessen disease severity for those already infected.

While a number of claims on efficacy of herbal remedies on COVID-19 have been made, to our knowledge none of such claims have gained on scientific basis for continued use or further research and development of the constituents into investigational products.

In Uganda, one of such herbal remedies is COVIDEX, this study therefore seeks to investigate the safety and efficacy of COVIDEX in the management of COVID-19.

DETAILED DESCRIPTION:
The SARS-CoV-2 pandemic continues to grow, with over 350,000 new infections and over 7,000 daily global deaths in May 2021 (WHO, 2021a). The current supplies of protective vaccines are too low to cover the worldwide demand hence researchers globally are urgently looking for interventions to prevent new infections, prevent disease progression, and lessen disease severity for those already infected. According to data released by the ministry of health, Uganda had 94,904 confirmed cases with 2752 deaths at the end of July 2021 (MoH, 2021). Fortunately, most of the cases confirmed had a mild illness for whom home-based symptomatic management with monitoring of clinical deterioration as per World Health Organization recommendations is sufficing (WHO, 2021b). However, despite providing symptomatic management, a therapeutic drug that would limit infection is greatly needed to stop COVID-19 disease progression. While a number of claims on efficacy of herbal remedies on COVID-19 have been made, to our knowledge none of such claims have gained on scientific basis for continued use or further research and development of the constituents into investigational products.

COVIDEX is a herbal formulation containing berberine as a primary anti-SARSCOV-2 compound notified by the Uganda National Drug Authority for supportive treatment in managing viral infections. Notably, this notification was done with a call for clinical trials to validate the claims of its anti-SARS COV-2 activity. This study therefore proposes to investigate the safety and efficacy of COVIDEXTm therapy in managing COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed/thumb printed and dated informed consent form
2. Willingness to comply with all study procedures and availability over the study duration
3. Patients aged 18years and above
4. Positive SARS-CoV-2 antigen rapid test and/or PCR positive for SARS-Cov-2 (COVID-19)
5. Symptomatic patients in the following categories; mild, moderate and severe: mild score 2 (limitation of activities), Moderately ill COVID-19 patients WHO score 3(Hospitalized with no oxygen therapy), which translates to moderately ill patients according to MOH Uganda, WHO Score 4 (Hospitalized with oxygen by mask or nasal prongs) and WHO score 5 (Non-invasive ventilation or high flow oxygen) which translates to severe COVID-19 disease on high flow oxygen patients according to the MOH Uganda COVID-19 disease category.

Exclusion Criteria:

1. Patients who report use of COVIDEX with-in three days prior to presentation to the hospital.
2. Clinical diagnosis of severe renal (defined by GFR ≤ 29 mL/min/1.73 m2) and hepatic impairment (defined by >2.5 times the upper normal value of ALT and AST).
3. Pregnancy or breast feeding.
4. Current use of remdesivir and molnupiravir therapy.
5. Active participation in another clinical trial or using another drug on compassionate use such as fluvoxamide.
6. Very ill patients with multiple comorbidities where determination of clinical outcome will be difficult as judged by the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety primary outcome | Daily for 30 days
  Incidence of severe adverse events of grade 3 and above Minimum score: 0, Maximum score: 4. The higher the score, the worse is the adverse event
Efficacy primary outcome: | Day 8
  Clinical recovery as measured by the WHO COVID ordinal improvement score Minimum score:0, Maximum score: 8. The higher the score, the worse is the clinical recovery

SECONDARY OUTCOMES:
SARS-CoV-2 antigen present in the nasopharynx | Day 8 and day 14
  SARS-CoV-2 antigen present in the nasopharynx
SARS-CoV-2 viral load in the nasopharynx as measured by the CT values | Day 8 and day 14
  SARS-CoV-2 viral load in the nasopharynx as measured by the CT values

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University Department of Pharmacology and Therapeutics, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided